CLINICAL TRIAL: NCT07202793
Title: Effectiveness and Tolerance of Respiratory Rehabilitation in Pulmonary Hypertension Associated With Chronic Obstructive Pulmonary Disease
Acronym: REHABTP
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Collaborators: Rehabilitation center, moulin vert (Unknown)
Responsible Party: Sponsor
Other Study IDs: REHABTP
Record Dates: First submitted 2025-08-04; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: COPD; Pulmonary Hypertension
Keywords: Rehabilitation; Pulmonary Disease; Chronic Obstructive; Pulmonary hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic obstructive pulmonary disease with pulmonary hypertension: Adults (≥18 years) who have spirometry-confirmed COPD and an intermediate or high echocardiographic probability of pulmonary hypertension, determined according to ESC/ERS criteria 1 year before or after rehabilitation ; completed ≥ 3 consecutive weeks of outpatient pulmonary rehabilitation (PR) at the University Hospital of Poitiers affiliated centre between 2013 and 2023
  ; performed a baseline and post-programme six-minute walk test (6MWT) under ATS guidelines.
- Chronic obstructive pulmonary disease without pulmonary hypertension: Adults (≥18 years) who have spirometry-confirmed COPD and no echocardiographic suspicion of pulmonary hypertension or low probability, determined according to ESC/ERS criteria 1 year before or after rehabilitation ; completed ≥ 3 consecutive weeks of outpatient pulmonary rehabilitation (PR) at the University Hospital of Poitiers affiliated centre between 2013 and 2023
  ; performed a baseline and post-programme six-minute walk test (6MWT) under ATS guidelines.

SUMMARY:
Observational study summary The goal of this observational study is to determine whether an outpatient pulmonary rehabilitation (PR) program-already known to be effective and safe for chronic obstructive pulmonary disease (COPD)-is equally effective and well-tolerated when COPD is complicated by pulmonary hypertension (PH).

Main question In adults with COPD + PH, does outpatient PR improve six-minute walk distance (6MWD) and remain safe, to the same extent as in adults with COPD without PH?

How the study is conducted

Researchers retrospectively analyse medical records from the University Hospital of Poitiers covering a ten-year period. Eligible participants are adults with COPD who completed at least three weeks of supervised PR and underwent echocardiography to assess PH probability. Two cohorts are compared:

COPD + PH (intermediate or high echocardiographic suspicion) COPD without PH (no echocardiographic suspicion) Key data collected Change in 6MWD between the start and end of PR (primary endpoint) Proportion of participants achieving a clinically meaningful improvement in 6MWD Occurrence of severe exacerbations (hospital- or emergency-treated events) during the year after PR All-cause mortality within one year Adverse events or program interruptions indicating PR tolerance

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Spirometry-confirmed chronic obstructive pulmonary disease with a post-bronchodilator FEV1 / FVC ratio below 0 .70
* Completion of at least three consecutive weeks of outpatient pulmonary rehabilitation between January 2013 and December 2023 at the University - Hospital of Poitiers centre
* Six-minute walk test performed within seven days before programme start and repeated during the final week
* Transthoracic echocardiogram carried out within one year before or one year after programme start, used to grade pulmonary hypertension

Exclusion Criteria:

* Pulmonary rehabilitation shorter than three weeks or missing six-minute walk test or echocardiogram data
* Chronic lung disease other than chronic obstructive pulmonary disease or previous lung transplantation

  -,Hospital admission for an acute chronic obstructive pulmonary disease exacerbation in the four weeks preceding rehabilitation
* Unstable cardiovascular disease that contraindicates exercise training
* Active cancer with an expected survival under one year
* Pregnancy at the time of rehabilitation
* Documented refusal to allow medical data to be used for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population consists of adults (18 years and older) with spirometry-confirmed chronic obstructive pulmonary disease who attended at least three consecutive weeks of supervised outpatient pulmonary rehabilitation at the University Hospital of Poitiers (France) between January 2013 and December 2023. Every individual had a six-minute walk test recorded both immediately before the programme and during its final week, plus a transthoracic echocardiogram performed within one year before or after programme start to grade the probability of pulmonary hypertension. Most candidates were current or former smokers with moderate-to-severe airflow limitation and common cardiometabolic or sleep-related comorbidities. Patients are classified into two analytic cohorts-COPD with pulmonary hypertension and COPD without pulmonary hypertension-according to their echocardiographic findings.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in six-minute walk distance (6MWD) | Up to 3 weeks
  Absolute difference (metres) between the 6-minute walk test performed at the start of the pulmonary-rehabilitation (PR) programme and the test repeated at the final session, following ATS/ACCP standards

SECONDARY OUTCOMES:
Participants achieving the minimum clinically important difference (MCID) in 6MWD | Up to 3 weeks
  Number and proportion of participants whose 6MWD rises by ≥ 30.5 m between baseline and the end of PR, the accepted MCID for this test
Severe COPD exacerbations | Between 0 and 12 months after PR
  Count of exacerbations requiring an emergency-department visit or hospital admission in the 12 months following completion of PR
All-cause mortality | Between 0 and 12 months after PR
  Death from any cause, confirmed through the French national death registry
Tolerance of PR | Day 1 and up to 3 weeks
  Number of adverse events occurring during the PR course or Number of programme interruptions due to acute causes (e.g., infection, exacerbation)

OTHER OUTCOMES:
Descriptive baseline data and course characteristics | Baseline
  Age, sex, BMI, smoking status, comorbidities; PR duration, reasons for any interruption; minimal SpO₂ recorded during each 6MWT; lung-function and echocardiographic variables

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Marie EMJ Jutant, MD PhD, Study Chair — CHU de Poitiers, University of Poitiers, France; Christian CG GIFFA, MD, Principal Investigator — CHU de Poitiers, University of Poitiers, France
Locations (1):
- CHU de Poitiers, University of Poitiers, France, Poitiers, Vienne, France

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared because this is a retrospective single-center study based on medical records, and no explicit consent for data sharing was obtained from participants.